CLINICAL TRIAL: NCT03213873
Title: Effects of the HiBalance-program: Linking Clinical Signs and Symptoms to Changes in the Brain in People With Parkinson´s Disease
Brief Title: Neuroplasticity in Parkinson´s Disease After Training
Acronym: BETA-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Erika Franzén, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2872/2016
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Physical Activity; Gait Disorders, Neurologic; Neural Degeneration
Keywords: Balance control; Exercise; Magnetic Resonance Imaging; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Gait Disorders, Neurologic; Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessors are masked to group allocation at baseline assessment. Care providers are masked to results of the assessments.
  Participants are masked to the studied intervention/treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HiBalance (Experimental): The HiBalance program is based on scientifically well-established principles of exercise training and postural control as well as current research on training in PD. The training will be conducted as a progressive individually adjusted group program in order to challenge the specific balance disorder of every participant and endorse progression. The intervention will be performed for an hour, 2 times/week in groups of six to eight participants for a total of 10 weeks and one home training session on their own.
  Interventions: Behavioral: HiBalance
- Speech therapy (Active Comparator): The control group will receive a group treatment (2 times/w for 10 w + 1 home training session) consisting of speech and communication therapy performed by a speech therapist. This intervention will be performed in a sitting position. The speech and communication treatment will aim at increasing vocal loudness and improving articulatory precision. Level of difficulty is gradually increased by progressing from using loud voice and clear speech in short and automatized utterances, to using the same technique in more complex sentences and situations. The group format is used to practice techniques in communicative situations and also to introduce increasing level of multitasking by combining speech training with cognitively more challenging tasks in the group training.
  Interventions: Behavioral: Speech and communication therapy

INTERVENTIONS:
Behavioral: HiBalance — Intervention of highly challenging balance training for 10 weeks.
  Arms: HiBalance
Behavioral: Speech and communication therapy — Intervention conducted by speech and language therapist for 10 weeks.
  Arms: Speech therapy

SUMMARY:
This project aims to determine the effects of the HiBalance program on neuroplastic changes in people with mild to moderate Parkinson´s disease. The main hypothesis is that highly challenging exercise will lead to greater gait and balance ability, increased levels of physical activity and an improved health related quality of life. The investigators further hypothesize that neuroplasticity changes will be seen in corresponding areas of the brain, neuropsychological changes on cognitive test measures, and that exercise will inhibit the degeneration of dopaminergic neurons in the brain through the mediation of neurotrophic factors.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disease affecting many physiological systems essential for balance control. New findings suggest that intensive, challenging and cognitively demanding exercises could induce neuroplasticity in PD. A new balance training (the HiBalance program) have therefore been developed; emphasizing critical aspects of balance control through highly challenging and progressive exercises incorporating dual/multi-tasking (Conradsson et al, 2012). In an RCT, the HiBalance-program was shown to improve balance, gait and physical activity level in favor for the training group (Conradsson et al, 2015). In this proposal the investigators will combine physiotherapy, neurology and neuroimaging to characterise and determine the effects on physical and cognitive symptoms as well as structural and functional changes and wet biomarkers in the brain after the training.

Participants will be recruited through Karolinska University Hospital and via announcements in relevant forums like for instance the Swedish Parkinson Association. According to earlier power calculations for detecting effects in balance and gait measures after this particular intervention, the investigators anticipate 40 to 50 participants in each group to detect significant changes.

The investigators will perform both per protocol analysis and intention to treat analysis using mixed model or repeated measurement ANOVAs if the data is normally distributed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson´s disease
* Hoehn & Yahr 2-3
* ≥ 60 years of age
* Be able to ambulate indoors without mobility aid
* Balance impairment

Exclusion Criteria:

* =< 21 points on MoCA
* Other medical conditions that could substantially influence balance performance, voice or speech performance or participation in the interventions
* Participating in an intensive exercise program for balance or speech during the last six months.

Additional exclusion criteria for the brain imaging will include the presence of; pacemakers, deep brain stimulators or other MRI incompatible implants, claustrophobia, inability to hear instructions without hearing aid, unilateral or bilateral blindness, severe diplopia, tremor, dyskinesia or dystonia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Eriksdotter, Professor, Study Chair — Karolinska Institutet, NVS department
Locations (1):
- Karolinska institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No
Currently we do not have IRB for sharing.

REFERENCES:
- [Background] Conradsson D, Lofgren N, Stahle A, Hagstromer M, Franzen E. A novel conceptual framework for balance training in Parkinson's disease-study protocol for a randomised controlled trial. BMC Neurol. 2012 Sep 27;12:111. doi: 10.1186/1471-2377-12-111. PMID 23017069
- [Background] Conradsson D, Lofgren N, Nero H, Hagstromer M, Stahle A, Lokk J, Franzen E. The Effects of Highly Challenging Balance Training in Elderly With Parkinson's Disease: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Oct;29(9):827-36. doi: 10.1177/1545968314567150. Epub 2015 Jan 21. PMID 25608520
- [Background] Franzen E, Johansson H, Freidle M, Ekman U, Wallen MB, Schalling E, Lebedev A, Lovden M, Holmin S, Svenningsson P, Hagstromer M. The EXPANd trial: effects of exercise and exploring neuroplastic changes in people with Parkinson's disease: a study protocol for a double-blinded randomized controlled trial. BMC Neurol. 2019 Nov 12;19(1):280. doi: 10.1186/s12883-019-1520-2. PMID 31718583
- [Background] Johansson H, Freidle M, Ekman U, Schalling E, Leavy B, Svenningsson P, Hagstromer M, Franzen E. Feasibility Aspects of Exploring Exercise-Induced Neuroplasticity in Parkinson's Disease: A Pilot Randomized Controlled Trial. Parkinsons Dis. 2020 Mar 25;2020:2410863. doi: 10.1155/2020/2410863. eCollection 2020. PMID 32300475
- [Derived] Steurer H, Gustafsson JK, Franzen E, Schalling E. Auditory-Perceptual Analysis of Speech Outcomes Following HiCommunication Intervention in Parkinson's Disease-A Secondary Analysis of a Randomized Controlled Trial. J Voice. 2025 Jul 8:S0892-1997(25)00234-6. doi: 10.1016/j.jvoice.2025.06.015. Online ahead of print. PMID 40628546
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Freidle M, Johansson H, Ekman U, Lebedev AV, Schalling E, Thompson WH, Svenningsson P, Lovden M, Abney A, Albrecht F, Steurer H, Leavy B, Holmin S, Hagstromer M, Franzen E. Behavioural and neuroplastic effects of a double-blind randomised controlled balance exercise trial in people with Parkinson's disease. NPJ Parkinsons Dis. 2022 Jan 21;8(1):12. doi: 10.1038/s41531-021-00269-5. PMID 35064138
- [Derived] Leavy B, Hagstromer M, Conradsson DM, Franzen E. Physical Activity and Perceived Health in People With Parkinson Disease During the First Wave of Covid-19 Pandemic: A Cross-sectional Study From Sweden. J Neurol Phys Ther. 2021 Oct 1;45(4):266-272. doi: 10.1097/NPT.0000000000000372. PMID 34369451
- [Derived] Johansson H, Ekman U, Rennie L, Peterson DS, Leavy B, Franzen E. Dual-Task Effects During a Motor-Cognitive Task in Parkinson's Disease: Patterns of Prioritization and the Influence of Cognitive Status. Neurorehabil Neural Repair. 2021 Apr;35(4):356-366. doi: 10.1177/1545968321999053. Epub 2021 Mar 10. PMID 33719728

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HiBalance | Speech Therapy
Started | 48 | 47
Completed | 40 | 35
Not Completed | 8 | 12
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Diagnosed w atypical PD after randomization | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HiBalance | Speech Therapy | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (5.9) | 71.1 (6.3) | 71.1 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 30 | 30 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 48 | 47 | 95
Disease stage Hoehn & Yahr [Count of Participants; unit: Participants] — Hoehn & Yahr stages (stage1 to 5) were clinically assessed with the guidance from MDS-UPDRS. Stage 2 is has less PD involvement than stage 3
  Hoehn Yahr Stage 2 =Bilateral or midline involvement without impairment of balance, Hoehn Yahr Stage 3 =Bilateral disease: mild to moderate disability with impaired postural reflexes; physically independent.
  Participants
    Hoehn Yahr Stage 2 | 39 | 34 | 73
    Hoehn Yahr Stage 3 | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mini-BESTest
Description: Mini-Balance Evaluation Systems Test a rating scale for dynamic balance incorporating 14 different balance and gait items that were assessed by a physical therapist on a scale from 0-2. Maximum points 28.
  0-28 points with higher scores indicating better balance control
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Population: All participants randomised included using intention-to-treat-analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
score on a scale
  Pre, observed values | 20.7 (3.4) | 21.0 (3.5)
  Post, observed values | 22.1 (3.0) | 21.8 (3.1)
Statistical Analysis 1: Comparison: HiBalance vs Speech Therapy; Test type: Superiority; p = 0.57, Mixed Models Analysis; Interaction effect time x group = 0.4, 95% CI 2-sided [-1.0 to 1.9]

2. Secondary Outcome: Gait Parameters
Description: Gait speed in m/sec
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Population: All participants randomised were included using intention-to-treat analyses.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
m/sec
  Pre, observed values | 1.2 (0.2) | 1.2 (0.2)
  Post, observed values | 1.3 (0.2) | 1.2 (0.2)
Statistical Analysis 1: Comparison: HiBalance vs Speech Therapy; Test type: Superiority; p = 0.25, Mixed Models Analysis; Interaction effect time x group = 0.05, 95% CI 2-sided [-0.03 to 0.12]

3. Secondary Outcome: Neuropsychological Tests
Description: Composite measure of executive functions of four tests:
  1. letter fluency
  2. the verbal fluency test: category switching
  3. the colour-word interference test: switch condition (Test 1, 2 and 3 from the Delis-Kaplan Executive Function System)
  4. the digit span total score (from Wechsler Adult Intelligence Scale)
  First, the scores of each of the four tests were standardised into z-scores using pre-scores. Models using different test were compared. The model including all four tests and using the robust diagonally weighted least square estimation was chosen based on fit values. Factor loadings of the model: verbal fluency = 1.000, the verbal fluency test: category switching= 0.887, the colour-word interference test: switch condition= -0.855, the digit span total score= 0.813. Last, the z-scores of each test and person were multiplied with the factor loadings and added together to create a sum score for each person and time point. A higher value = greater executive functions
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Measure: Mean (Standard Deviation); unit: z-scores
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
z-scores
  Pre, observed values | 0.6 (2.6) | -0.7 (2.4)
  Post, observed values | 1.5 (2.6) | 0.1 (3.0)
Statistical Analysis 1: Comparison: HiBalance vs Speech Therapy; Test type: Superiority; p = 0.75, Mixed Models Analysis; Interaction effect time x group = 0.2, 95% CI 2-sided [-0.8 to 1.1]

4. Secondary Outcome: Quality of Life Questionnaires
Description: The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living (mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communications and bodily discomfort).
  The sum score is as a percentage score ranging between 0 and 100. Higher is better
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
score on a scale
  Pre, observed values | 19.7 [13.1 to 30.9] | 17.8 [9.8 to 27.7]
  Post, observed values | 17.5 [7.3 to 23.0] | 11.9 [7.3 to 25.4]

5. Secondary Outcome: Movement Disorder Society - Unified Parkinsons Disease Rating Scale (MDS-UPDRS)
Description: Disease severity/symtoms in Parkinson's disease, Movement Disorder Society - Unified Parkinsons disease rating scale (MDS-UPDRS) Total score.
  Higher score is worse, ranging from 0-272
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
score on a scale
  Pre, observed values | 51.0 (18.8) | 50.4 (15.5)
  Post, observed values | 48.2 (17.8) | 45.8 (16.8)

6. Secondary Outcome: Physical Activity Measured With Accelerometers
Description: Number of Steps per day.
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Measure: Median (Inter-Quartile Range); unit: steps per day
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
steps per day
  Pre, observed values | 4936.6 [3250.1 to 6798.9] | 5462.4 [3094.6 to 7785.4]
  Post, observed values | 4800.8 [2839.1 to 6470.1] | 5609.5 [4048.0 to 8628.9]

7. Secondary Outcome: Structural Magnetic Resonance Imaging
Description: Intervention dependent changes in brain structure i.e. gray matter volume measured as voxels Analyses defined as: were there any significant clusters of voxels explained by the interaction of group and time. In other words, were there significant changes in voxel activity that depended on the interventions when using a cluster-based threshold using group statistics..
  Note that it is not possible to report this outcome per group. Additionally, MR statistics are not reported as measures of central tendency such as the mean or any alternatives provided.
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Measure: Number; unit: Significant clusters of voxels
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 34 | 31
Significant clusters of voxels | 0 | 0

8. Secondary Outcome: Task-induced Brain Activity as Measured by Functional Magnetic Resonance Imaging
Description: Intervention dependent changes in task-induced brain activity, voxel-wise analyses of whole brain. (Name of the task performed during fMRI; the serial reaction time task.)
  Analyses defined as: were there any significant clusters of voxels explained by the interaction of group and time. In other words, were there significant changes in voxel activity that depended on the interventions when using a cluster-based threshold. The measure type number was chosen because we estimated the number of significant clusters of voxels. Group statistics were perfromed
  Note that for task fMRI interaction analyses, there are no meaningful values to report for the groups respectively.
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Population: All participants without missing or too low-quality fMRI data were included
Measure: Number; unit: significant clusters of voxels
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 32 | 28
significant clusters of voxels | 0 | 0

9. Secondary Outcome: Wet Biomarkers
Description: Mature Brain-derived neurotrophic factor (mBDNF) in serum
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
pg/mL
  Pre, observed values | 38010.8 (7956.7) | 37805.3 (5928.3)
  Post, observed values | 37169.4 (8044.6) | 35945.8 (6208.5)

10. Other Pre Specified Outcome: Dysarthria
Description: The Dysarthria Assessment also includes the Questionnaire on Acquired Speech Disorders (QASD, Swedish: Självsvarsformulär om Förvärvade Talstörningar) which is a self-report instrument that captures the subjective symptoms and experiences of individuals living with acquired speech disorders. Three subscales are included: "My Speech and Language", "Speech and Language in Social Interaction", and "Personal and Environmental Factors". Each item is rated on a four-point scale from 0 (definitely false) to 3 (definitely true), with higher scores indicating more severe symptoms. The overall QASD score was determined by calculating the average score of all sub-scales.
Time Frame: Pre intervention baseline
Population: This variable were never analysed pre and post since it is not sensitive in patients with mild dysarthria. The variable was just used for describing the group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 47 | 43
score on a scale | 0.66 (0.44) | 0.43 (0.35)

11. Other Pre Specified Outcome: Voice Strength
Description: The recordings were performed according to standardised routines for high-quality recordings in a sound-proof recording studio with the equipment Sony Digital Audio Tape Deck DTC-ZE700 and the software Sopran (version 1.0.22 © Tolvan Data). Measures were performed by a speech and language pathologist.
  The outcome measure from the studio recordings used in the present study was mean voice sound level (dB SPL) in reading a Swedish standardised text.
Time Frame: Pre intervention baseline and post intervention at 10 weeks
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | HiBalance | Speech Therapy
Number analyzed (Participants) | 48 | 47
dB
  Pre, observed values | 70.3 (3.5) | 70.8 (4.0)
  Post, observed values | 70.6 (3.9) | 73.0 (4.0)

ADVERSE EVENTS:
Time Frame: During the 10 weeks of the interventions.
Arm/Group | HiBalance | Speech Therapy
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 8/48 | 0/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HiBalance (N=48) | Speech Therapy (N=47)
Non-injurious falls (Musculoskeletal and connective tissue disorders) | 7 | 0
Calf-muscle strain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT03213873/Prot_SAP_000.pdf